CLINICAL TRIAL: NCT01913184
Title: EFFECT OF DRUG TARGETING NEBULIZATION ON LUNG DELIVERY
Brief Title: Lung Bioavailability With Continuous or Discontinuous Nebulization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AKITA continuous
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Continuous nebulization (Active Comparator): Continuous nebulization with AKITA
  Interventions: Device: AKITA
- Discontinuous nebulization (Experimental): Discontinuous nebulization with AKITA
  Interventions: Device: AKITA

INTERVENTIONS:
Device: AKITA

SUMMARY:
To compare the continuous and sicontinuous delivery of drug with AKITA.

ELIGIBILITY:
Inclusion Criteria:

* no lung disease
* no allergy

Exclusion Criteria:

* smoker

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Lung bioavailability by urinary monitoring | 24h after the nebulization

SECONDARY OUTCOMES:
Duration of the nebulization | After the nebulization

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Reychler G, Aubriot AS, Masquelier J, Muccioli GG, Liistro G. Effect of drug-targeting nebulization on lung delivery. Arch Bronconeumol. 2014 Nov;50(11):500-1. doi: 10.1016/j.arbres.2013.10.014. Epub 2013 Dec 29. No abstract available. English, Spanish. PMID 24380752